CLINICAL TRIAL: NCT07339878
Title: Criteria for Selecting First-line Metastatic Treatment for Patients With Urothelial Carcinoma: Observational, Multicenter, Real-world Study
Brief Title: Criteria for Selecting First-line Metastatic Treatment for Patients With Urothelial Carcinoma
Acronym: FLORAL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9770
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Urothelial Carcinoma
Keywords: Urothelial Carcinoma; Enfortumab Vedotin; Pembrolizumab
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The standard first-line treatment for metastatic urothelial carcinoma has become the combination of Enfortumab Vedotin and Pembrolizumab following the publication of the EV-302 study results at the end of 2024. Another standard remains in 2025 for patients who are not eligible for the EV Pembrolizumab combination, namely platinum-based chemotherapy +/- avelumab in cases of non-progression. The objective of the FLORAL study is to determine the characteristics of these patients and the reasons that led clinicians to prefer a first-line treatment based on platinum salts.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Metastatic urothelial carcinoma
* Treated with first-line metastatic therapy since October 2024

Exclusion Criteria:

* Patient who expressed opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adut atient with metastatic urothelial carcinoma and reated with first-line metastatic therapy since October 2024
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Description of the clinical characteristics of patients recently treated with first-line metastatic therapy for urothelial carcinoma | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service Oncologie Médicale - CHU de Strasbourg - France, Strasbourg, France